CLINICAL TRIAL: NCT00760344
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate Treatment With SYR-472 in Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of SYR-472 in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-06-TL-SYR-472-006; U1111-1129-7916 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — trelagliptin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- SYR-472 3.125 mg QD (Experimental): (with lifestyle modification and/or metformin stable dose therapy)
  Interventions: Drug: SYR-472
- SYR-472 12.5 mg QD (Experimental): (with lifestyle modification and/or metformin stable dose therapy)
  Interventions: Drug: SYR-472
- SYR-472 50 mg QD (Experimental): (with lifestyle modification and/or metformin stable dose therapy)
  Interventions: Drug: SYR-472
- SYR-472 100 mg QD (Experimental): (with lifestyle modification and/or metformin stable dose therapy)
  Interventions: Drug: SYR-472
- Placebo QD (Placebo Comparator): (with lifestyle modification and/or metformin stable dose therapy)
  Interventions: Drug: Placebo
- Sitagliptin 100 mg QD (Active Comparator): (with lifestyle modification and/or metformin stable dose therapy)
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: SYR-472 — SYR-472 3.125 mg, tablets, orally, once daily with lifestyle modification and/or metformin stable dose therapy for up to 12 weeks.
  Arms: SYR-472 3.125 mg QD
Drug: SYR-472 — SYR-472 12.5 mg, tablets, orally, once daily with lifestyle modification and/or metformin stable dose therapy for up to 12 weeks.
  Arms: SYR-472 12.5 mg QD
Drug: SYR-472 — SYR-472 50 mg, tablets, orally, once daily with lifestyle modification and/or metformin stable dose therapy for up to 12 weeks.
  Arms: SYR-472 50 mg QD
Drug: SYR-472 — SYR-472 100 mg, tablets, orally, once daily with lifestyle modification and/or metformin stable dose therapy for up to 12 weeks.
  Arms: SYR-472 100 mg QD
Drug: Placebo — SYR-472 placebo-matching tablets, orally, once daily with lifestyle modification and/or metformin therapy for up to 12 weeks.
  Arms: Placebo QD
Drug: Sitagliptin — Sitagliptin 100 mg, tablets, orally, once daily with lifestyle modification and/or metformin stable dose therapy for up to 12 weeks.
  Other Names: Januvia™
  Arms: Sitagliptin 100 mg QD

SUMMARY:
The purpose of this study is to determine the efficacy and safety of SYR-472, once daily (QD), in subjects with type 2 diabetes mellitus who have not achieved glycemic control with diet and exercise, or by taking metformin.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is a complex metabolic disorder characterized by abnormal insulin secretion and glucose homeostasis, resulting from impaired pancreatic beta-cell function and insulin resistance in target tissues. The worldwide prevalence of type 2 diabetes mellitus is reaching epidemic proportions, and the total number of cases is expected to reach 221 million by 2010. The high incidence of the disease and its associated complications places a significant burden on healthcare systems.

The primary risk factor for the development of type 2 diabetes mellitus is obesity and its associated insulin resistance. Insulin resistance is characterized by an impaired response to the physiologic effects of insulin and leads to decreased cellular glucose uptake, increased hepatic gluconeogenesis, and a compensatory increase in insulin secretion that contributes to beta-cell exhaustion. Therefore in the insulin-resistant state, blood glucose and insulin levels are increased. The relationship between improved glycemic control in patients with type 2 diabetes mellitus and the delay or prevention of comorbidities has been reported in the Diabetes Control and Complications Trial and the United Kingdom Prospective Diabetes Study. Therefore, reduction of persistent hyperglycemia is the highest priority in treating this disease.

Diet and exercise are important and effective measures for maintaining glycemic control in individuals with insulin resistance, impaired glucose tolerance, and type 2 diabetes mellitus, particularly in the early stages of disease progression. In cases where diet and exercise alone fail to adequately maintain glycemic control, oral antidiabetic drugs are typically used. Combination oral therapy and eventually insulin are usually required to maintain lower blood glucose levels but can result in adverse effects including hypoglycemia and weight gain. Therefore, novel safe and effective antidiabetic therapies are needed.

Dipeptidyl peptidase-4 is a ubiquitous aminopeptidase that is widely expressed in many tissues; it is thought to be primarily responsible for the in vivo degradation of at least two gut-derived incretin hormones, namely glucagon-like peptide-1 and glucose-dependent insulinotropic peptide, which are both released in response to nutrient ingestion. Glucagon-like peptide-1 has been demonstrated to augment glucose-dependent insulin secretion; suppress glucagon release and hepatic gluconeogenesis; inhibit gastric emptying, and reduce appetite and food intake. Glucagon-like peptide-1 and glucose-dependent insulinotropic peptide also have been shown to promote insulin biosynthesis and stimulate beta cell proliferation and survival. Orally available inhibitors of dipeptidyl peptidase-4 activity have been developed that increase intact postprandial glucagon-like peptide-1 levels after oral administration.

SYR-472 is a selective inhibitor of dipeptidyl peptidase-4 in development to improve glycemic control in patients with type 2 diabetes mellitus. The aim of this study is to evaluate SYR-472 in subjects with type 2 diabetes mellitus who have not previously achieved adequate glycemic control with lifestyle modification (diet/exercise) or metformin antidiabetic monotherapy. Study participation is anticipated to be up to 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Had a historical diagnosis of type 2 diabetes mellitus.
* Had undergone less than 7 days of any antidiabetic therapy except lifestyle modification (diet/exercise) within 8 weeks prior to Screening; or has received metformin monotherapy for at least 8 weeks prior to Screening and maintained a stable daily dose of metformin for at least 12 weeks prior to randomization.
* If receiving metformin monotherapy at randomization must have been at least 75% compliant with his or her regimen during the Run in/Stabilization Period as determined by subject diary and investigator assessment.
* Had received no treatment with antidiabetic agents other than metformin within the 8 weeks prior to Screening.
* The subject has an glycosylated hemoglobin concentration between 7.0% and 10.0%, inclusive, at Screening and at the Week -1 Visit.
* Had a body mass index between 23 and 45 kg/m2.
* A C-peptide concentration is greater than or equal to 0.8 ng/mL (greater than or equal to 0.26 nmol/L).
* A fasting plasma glucose concentration is less than 275 mg/dL (less than 15.27 mmol/L) at Screening and at the Week -1 Visit.
* If the subject regularly uses other non-excluded medications, he or she must be on a stable dose for at least the 4 weeks prior to Screening.
* The subject has a systolic blood pressure reading of less than 160 mm Hg and a diastolic pressure reading of less than 100 mm Hg.
* The subject has a hemoglobin value greater than or equal to 12 g/dL (greater than or equal to 120 g/L) for men and greater than or equal to 10 g/dL (greater than or equal to 100 g/L) for women.
* Had an alanine aminotransferase level is less than or equal to 3 times the upper limit of normal.
* A male subject has a serum creatinine value of less than 1.5 mg/dL (less than 133 μmol/L); a female subject has a serum creatinine value of less than 1.4 mg/dL (less than 124 μmol/L).
* Had a urine albumin/creatinine ratio of less than 1000 μg/mg at Screening.
* Had a thyroid-stimulating hormone level less than or equal to the upper limit of the normal range and the subject is clinically euthyroid.
* A female subject of childbearing potential who is sexually active must agree to use adequate contraception, and must be neither pregnant nor lactating from Screening and throughout the duration of the study.
* Was able and willing to monitor his or her own blood glucose concentrations with a home glucose monitor.
* Had no major illness or debility that in the investigator's opinion prohibits the subject from completing the study.

Exclusion Criteria:

* Was being concurrently treated with antidiabetic therapy other than metformin and lifestyle intervention.
* Had a history of cancer, other than squamous cell or basal cell carcinoma of the skin that has not been in full remission for at least 5 years prior to Screening.
* Had a history of laser treatment for proliferative diabetic retinopathy within the 6 months prior to Screening.
* Had a history of treated diabetic gastric paresis.
* Had a New York Heart Association class III or IV heart failure regardless of therapy.
* Had a history of coronary angioplasty, coronary stent placement or coronary bypass surgery, myocardial infarction, or stroke within the 6 months prior to Screening.
* Had a history of hemoglobinopathy that may affect determination of glycosylated hemoglobin.
* Had a history of infection with human immunodeficiency virus.
* Had a history of a psychiatric disorder that in the investigator's opinion will affect the subject's ability to participate in the study.
* Had a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) or substance abuse (defined as illicit drug use) within the 2 years prior to Screening.
* Was required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Ingested or received systemically injected glucocorticoids within the 3 months prior to randomization.
  * Used prescription or over-the-counter weight-loss drugs within the 3 months prior to randomization.
  * Received any investigational drug within the 30 days prior to Screening or has received an investigational antidiabetic drug within the 3 months prior to Screening.
* Had received previous treatment in an investigational study of SYR-472.
* Had a known hypersensitivity to any compound related to SYR-472 or Sitagliptin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glycosylated hemoglobin | Week 12 or Final Visit

SECONDARY OUTCOMES:
Change from baseline in glycosylated hemoglobin | Weeks 4, 8 and 12 or Final Visit.
Change from baseline in fasting plasma glucose | Weeks 1, 2, 4, 8, and 12 or Final Visit
Change from baseline in 1,5-Anhydroglucitol | Weeks 2, 4, 8, and 12 or Final Visit.
Change from baseline in Proinsulin | Weeks 4, 8, and 12 or Final Visit.
Change from baseline in Insulin | Weeks 4, 8, and 12 or Final Visit.
Change from baseline in Proinsulin/insulin ratio | Weeks 4, 8, and 12 or Final Visit.
Change from baseline in C-peptide | Weeks 4, 8, and 12 or Final Visit.
Change from baseline in Homeostasis model assessment of insulin resistance. | Weeks: 4, 8, and 12 or Final Visit.
Change from baseline in Homeostasis model assessment of beta-cell function. | Weeks 4, 8, and 12 or Final Visit.
Incidence of marked hyperglycemia (fasting plasma glucose greater than or equal to 200 mg/dL [11.10 mmol/L]). | Weeks 4, 8 and 12 or Final Visit.
Incidence of rescue. | Weeks 1, 2, 4, 8, and 12 or Final Visit.
Clinical response endpoint incidence of glycosylated hemoglobin less than or equal to 6.5%. | Week 12 or Final Visit
Clinical response endpoint incidence of glycosylated hemoglobin less than or equal to 7.0%. | Week 12 or Final Visit
Change from baseline in Fasting lipids (triglycerides, total cholesterol, high-density lipoprotein cholesterol and low-density lipoprotein cholesterol). | Weeks 4, 8, and 12 or Final Visit.
Body weight. | Weeks 4, 8, and 12 or Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda
Locations (112):
- United States (105):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Phoenix, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Anderson, Arkansas
  - Little Rock, Arkansas
  - Pine Bluff, Arkansas
  - Carmichael, California
  - Chino, California
  - Long Beach, California
  - Los Angeles, California
  - Los Gatos, California
  - Orange, California
  - Pico Rivera, California
  - Rolling Hills Estates, California
  - Roseville, California
  - Rowland Heights, California
  - Sacramento, California
  - Santa Ana, California
  - Stockton, California
  - Torrance, California
  - Arvada, Colorado
  - Colorado Springs, Colorado
  - Highlands Ranch, Colorado
  - Avon, Connecticut
  - Rocky Hill, Connecticut
  - Newark, Delaware
  - Aventura, Florida
  - Edgewater, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Merritt Island, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Zanesville, Florida
  - Atlanta, Georgia
  - Roswell, Georgia
  - Waycross, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Avon, Indiana
  - Fort Wayne, Indiana
  - Des Moines, Iowa
  - Waterloo, Iowa
  - Topeka, Kansas
  - Wichita, Kansas
  - Crestview, Kentucky
  - Oxon Hill, Maryland
  - Detroit, Michigan
  - Troy, Michigan
  - Olive Branch, Mississippi
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - West Caldwell, New Jersey
  - Wildwood Crest, New Jersey
  - Albuquerque, New Mexico
  - East Islip, New York
  - Lewiston, New York
  - New York, New York
  - North Massapequa, New York
  - Wantagh, New York
  - Hickory, North Carolina
  - Statesville, North Carolina
  - Tabor City, North Carolina
  - Bismarck, North Dakota
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Mason, Ohio
  - Wadsworth, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Medford, Oregon
  - Bensalem, Pennsylvania
  - Connellsville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Shippensburg, Pennsylvania
  - Charleston, South Carolina
  - Greer, South Carolina
  - North Myrtle Beach, South Carolina
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - New Tazewell, Tennessee
  - Carrolton, Texas
  - Dallas, Texas
  - Georgetown, Texas
  - Houston, Texas
  - Killeen, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Spanish Fork, Utah
  - Richmond, Virginia
  - Suffolk, Virginia
  - Virginia Beach, Virginia
  - Spokane, Washington
- Mexico (7):
  - Zapopan, Jalisco
  - Monterrey, Nuevo León
  - Puebla City, Puebla
  - Mexico City
  - Monterrey
  - Nezahualcóyotl
  - Veracruz